CLINICAL TRIAL: NCT06640192
Title: Clinical Trial Phase II, Multicenter, Open-label, Randomized and Controlled Trial to Eliminate the Latent Reservoir of HIV-1 by Administering High Doses of Antiretroviral Drugs.
Brief Title: Administration of High Doses of Antiretroviral Drugs to Eliminate the Latent HIV-1 Reservoir
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOSAGE
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Triple therapy antiretroviral drugs on their usual regimen containing an integrase inhibitor
  Interventions: Drug: Standardised triple antiretroviral therapy
- Intervention (Experimental): High doses of triple therapy antiretroviral drugs: dolutegravir 50 mg/12 h, maraviroc 300 mg/12 h and lamivudine 300 mg/12 h.
  Interventions: Drug: High doses Triple therapy antiretroviral drugs

INTERVENTIONS:
Drug: Standardised triple antiretroviral therapy — patients have to use Triple therapy antiretroviral drugs on their usual regimen containing an integrase inhibitor. There are many types of drugs within this group, so they are not specified.
  Arms: Control
Drug: High doses Triple therapy antiretroviral drugs — dolutegravir 50 mg/12 h, maraviroc 300 mg/12 h and lamivudine 300 mg/12 h
  Arms: Intervention

SUMMARY:
The HIV epidemic represents one of the greatest health challenges worldwide, with important social and economic implications for public health. Although combination antiretroviral therapy (TAR) is effective in controlling infection and delaying disease onset, as well as improving the quality of life of infected persons, the relevant medical needs caused by HIV-1 infection are not yet fully met by TAR. The main obstacle to curing HIV is the establishment and maintenance of the viral reservoir. Therefore, we believe that this clinical trial will provide knowledge, for the first time, of the increase of antiretroviral drug levels in lymphatic tissue achieved by simultaneous administration of antiretroviral drugs at higher than usual doses, and their effect on persistent viral replication in intestinal lymphatic tissue and, as a consequence, on the latent cellular reservoir of HIV.

DETAILED DESCRIPTION:
Data on the penetration of antiretrovirals into the tissues of long-term treated HIV patients are very limited. Previous pharmacokinetic studies indicate that tissue concentrations of the drug are much lower than those observed in plasma of HIV-infected patients or healthy volunteers. In addition, another study has reported that intracellular levels of antiretrovirals are much lower in lymphoid tissues than in peripheral blood after 6 months of TAR initiation, and these levels correlated inversely with ongoing viral replication.

In the line of research that we are raising, a previous study has reported a decrease in intracellular HIV RNA in lymphoid tissue when dolutegravir was administered at higher than usual doses. This is an important advance and new studies should be implemented with a design that allows to potentiate this strategy and significantly decrease the size of the viral reservoir in tissues.

If the hypothesis of the project, which consists mainly in the reduction or elimination of the HIV reservoir, is demonstrated, there would be very important consequences in the area of functional cure of HIV and/or reduction of chronic persistent inflammation, which could generate changes in conventional treatment schemes with great scalability. In addition, it is possible that by decreasing levels of persistent viral replication, an improvement in levels of immune activation and inflammation may also be observed, which would contribute positively to the overall health of the patient. Oral antiretroviral medication is proposed in order to compound a three-drug antiretroviral regimen. The three antiretroviral drugs have been chosen because they are the only ones that allow administration at higher doses without causing increased toxicity: dolutegravir 50 mg/12 h, maraviroc 300 mg/12 h and lamivudine 300 mg/12 h.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, after receiving information about the study design, the aims of the study, the possible risks that may arise from it and the fact that they can refuse to collaborate at any time, give written consent to participate in the study.
* Be over 18 years of age and under 60 years of age.
* Understand the purpose of the study and be available to perform the visits and procedures established in the protocol.
* Persons with HIV being followed up in HIV consultations.
* Antiretroviral treatment with a triple regimen containing an integrase inhibitor.
* Undetectable plasma viral load (<50 copies of HIV RNA in blood plasma) for at least 12 months prior to inclusion.
* No history of prior virologic failure.
* No known gastrointestinal disease.
* R5 viral tropism, determined on proviral DNA.
* In women: negative urine pregnancy test performed within 7 days prior to the start of study treatment in women of childbearing age and if < 2 years post menopause.
* Women of childbearing age and male partners of childbearing age must agree to use a highly effective method of contraception (such as surgical sterilization, double barrier method, oral contraceptives, or hormonal contraceptive implants) and to continue using them until 6 months after the last dose of treatment.

Exclusion Criteria:

* Chronic Hepatitis B (HBsAg +)
* Untreated chronic hepatitis C
* Viral tropism X4
* Pregnancy or planning to become pregnant during the course of the study.
* Lactation.
* Abnormal coagulation parameters (PT> or equal to 1.2 LSN).
* Thrombocytopenia (platelet count <50000).
* Transaminases in values greater than 3 times normal.
* Impaired renal function (plasma creatinine >1.5 mg/dl, creatinine clearance <60 ml/min/1.73 m2).
* Contraindications for the performance of any of the study procedures (colonoscopy/bowel biopsy) or conscious sedation.
* Anemia (greater than or equal to grade 1).
* Administration of aspirin, ibuprofen, warfarin or other agents that interfere with the coagulation cascade are prohibited 1 week before endoscopy.
* Concomitant treatment with cytochrome CYP3A inducers or inhibitors.
* Patients in whom there is a contraindication for use according to the established in the technical data sheet or known hypersensitivity to the drugs under investigation or who, according to the investigator's criteria, it is not advisable to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the variation in the size of the latent cellular reservoir of HIV-1 in lymphoid tissue and peripheral blood after administration of high doses of antiretroviral drugs. | 48 weeks
  Latent cell reservoir size by measuring total and intact proviral DNA (IPDA).

SECONDARY OUTCOMES:
To evaluate the variation of intracellular HIV RNA in total CD4+ T cells and memory phenotypes from baseline to weeks 24 and 48 in both blood and lymphoid tissue. | 48 weeks
  HIV replication by measuring cell-associated HIV RNA (ca-HIV-RNA) and HIV RNA levels in blood and lymphoid tissue.
To compare changes in distribution and activation markers ( CD25, HLA-DR among others) in T-cell subpopulations (naïve and memory phenotypes). | 48 weeks
  Activation/inflammation markers (HLA-DR, CD25, among others) in blood and intestinal T-cell subpopulations.
To evaluate the effects of the intervention on markers of inflammation and bacterial translocation. | 48 weeks
  Levels of plasma biomarkers of activation/inflammation and bacterial translocation (IL-6, CRP, TNF, sCD14, among others).
To determine antiretroviral drug concentrations in blood and gastrointestinal tract tissue. | 48 weeks
  Antiretroviral drug concentrations in lymphoid tissue and peripheral blood.
To correlate markers of viral persistence (intact HIV DNA and ca-HIV RNA) with drug concentrations, as well as with activation and inflammation parameters of cell subpopulations and plasma. | 48 weeks
  Colonoscopy examination and collection of intestinal tissue samples (biopsy) for determination of viral reservoir variables (proviral DNA and intracellular HIV RNA) and antiretroviral drug levels.
Incidence of Adverse Events with experimental treatment regimen (Safety and Tolerability) | 48 weeks
  Incidence and types of adverse reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Moreno Guillen, Principal Investigator — IRYCIS. Hospital Universitario Ramón y Cajal. Madrid, Spain.
Locations (2):
- Spain (2):
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No